CLINICAL TRIAL: NCT05493722
Title: Optimization of Deep Brain Stimulation Parameters in Patients With Medically Refractory Epilepsy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: NEUROSURG-2021-29636
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Refractory Epilepsy; Deep Brain Stimulation
Keywords: Refractory Epilepsy; deep brain stimulation
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to a stimulation order at the baseline visit with optimized settings (OS) stimulation occurring for a total of 8 months and physician-selected settings (PS) stimulation chosen for a total of 4 months. For example, a patient may undergo PS setting stimulation from 4-8 months, then undergo OS setting stimulation from 8-12 and 12-16 months. Thus, there are three possible stimulation groups (1. PS, OS, OS; 2.OS, PS, OS; 3. OS, OS, PS).
Who Masked: Investigator, Outcomes Assessor
Masking Description: A study coordinator who is blinded to the chosen stimulation setting will check the data daily to ensure the patient is wearing the device properly and recording seizure events. At each optimization visit, the MoCA and QOLIE-10P surveys will also be administered to the participants by a member of the research team who is blinded to the group the participant is assigned to.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes

ARMS (3):
- Stimulation Group A (Experimental): Participants with already implanted DBS will receive stimulation order 1. PS, OS, OS.
  Interventions: Other: PS and OS stimulation order 1
- Stimulation Group B (Experimental): Participants with already implanted DBS will receive stimulation order 1. OS, PS, OS.
  Interventions: Other: PS and OS stimulation order 2
- Stimulation Group C (Experimental): Participants with already implanted DBS will receive stimulation order 1. OS, OS, PS.
  Interventions: Other: PS and OS stimulation order 3

INTERVENTIONS:
Other: PS and OS stimulation order 1 — PS, OS, OS
  Arms: Stimulation Group A
Other: PS and OS stimulation order 2 — OS, PS, OS
  Arms: Stimulation Group B
Other: PS and OS stimulation order 3 — OS, OS, PS
  Arms: Stimulation Group C

SUMMARY:
Deep brain stimulation (DBS) is used to treat epilepsy in cases where patients are medically refractory and are not candidates for surgical resection. This therapy has been shown to be effective in seizure reduction, yet very few patients achieve the ultimate goal of seizure freedom. Implantable neural stimulators (INSs) have many parameters that may be adjusted, and could be tuned to achieve very patient specific therapies. This study will develop a platform for stimulation setting optimization based on power spectral density (PSD) measures.

ELIGIBILITY:
Inclusion Criteria:

* medically refractory epilepsy
* already have a deep brain stimulator in place

Exclusion Criteria:

* severe dementia at investigator discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
Difference in broadband power with different settings | One year from baseline
  Different settings include different combinations of stimulation amplitude, frequency and pulse width. The full spectrum PSD data from all of the in-clinic recordings at all of the unique settings will be combined to look at the resulting difference in broadband power.
Difference in frequency band-specific low-frequency power (LFP) with different settings | One year from baseline
  Different settings include different combinations of stimulation amplitude, frequency and pulse width. The full spectrum PSD data from all of the in-clinic recordings at all of the unique settings will be combined to look at the resulting difference in frequency band-specific LFP.

SECONDARY OUTCOMES:
Identify all seizures | one year from baseline
  Detecting generalized tonic-clonic seizures using a wearable sensor wristband and patients-reported seizure activity.
Scores on Montreal Cognitive Assessment, MoCA | one year from baseline
  This is a brief cognitive assessment used to look at side effects of stimulation settings
Scores on epilepsy-specific quality of life questionnaire (QOLIE-10P) | One year from baseline
  This is a brief cognitive assessment used to look at side effects of stimulation settings

CONTACTS AND LOCATIONS:
Overall Officials: Robert McGovern, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States